CLINICAL TRIAL: NCT05048953
Title: The Relationship Between Changes in Thickness, Echogenicity and Fasciculation of Skeletal Muscle and Intensive Care Unit - Acquired Weakness
Brief Title: The Use of Musculoskeletal Ultrasound for the Detection of ICU-Acquired Weakness
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Collaborators: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Dr Sabin Bhandari, DM resident, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: IERB No 132(6-1)t2, 078/079
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: ICU Acquired Weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRC GROUP: All newly admitted patients (shifted to ICU within 48 h of hospital admission), aged ≥ 16 years and expected to stay in ICU or critical care areas for 7 days will be included in the study after excluding those who fulfill excluding criterial. In all the participants, muscle strength will be assessed at day 1, day 4 and day 7, if the patients are awake as assessed by Richmond Agitation Sedation Scale (RASS) (19) between -1 and 1, and cooperative (20) assessed by being able to follow at least 3 out of 5 verbal commands with facial muscles (scored by the Score of 5 Questions). Assessment will be done by an ICU physician blinded to the result of ultrasound. The MRC score will be used for assessment of strength in the following six muscle groups bilaterally: wrist dorsiflexors, elbow flexors, shoulder abductors, hip flexors, knee extensors and ankle dorsiflexors. ICU-AW will be defined as MRC sum score < 48, in accordance with the international consensus statement.(1)
  Interventions: Diagnostic Test: Muscle ultrasound measurements (the index test)
- Muscle ultrasound measurements (the index test): Muscle ultrasound will be performed by an ICU faculty or a DM resident of Critical care medicine (who has an experience of at least 25 muscle ultrasonography with at least 10 muscle ultrasonography performed under supervision) (21) and will be blinded to the result of MRC score of the patient. Muscle ultrasound images on day 1, day 4 and day 7 will be obtained in the participants.
  The following parameters will be measured by muscle ultrasound
  1. Muscle thickness
  2. Muscle echogenicity
  3. Muscle fasciculations Muscle thick

INTERVENTIONS:
Diagnostic Test: Muscle ultrasound measurements (the index test) — The following parameters will be measured by muscle ultrasound
  1. Muscle thickness
  2. Muscle echogenicity
  3. Muscle fasciculations
  Groups: MRC GROUP

SUMMARY:
Intensive Care Unit-Acquired Weakness (ICU-AW) is a clinical entity frequently encountered in critically ill patients that have both short term and long-term implications.

The current gold standard of diagnosis is by assessment of manual muscle strength, using the 6-grade Medical Research Council (MRC) sum score. However, not all Intensive Care Unit (ICU) admitted patients are conscious or cooperative enough to use MRC sum score for the diagnosis of ICU-AW. Ultrasound imaging of muscles has emerged as a valid and reliable tool for providing qualitative and quantitative details about muscle disease and has been suggested as an alternative to assess ICU-AW in critically ill patients in whom the MRC cannot be assessed. This study will be a prospective observational study to evaluate the relationship between the trend of changes in muscle thickness, echogenicity and fasciculations during the first 7 days of ICU stay as measured by ultrasound and ICU-AW among critically ill patients. The study will be performed in the ICU of TU Teaching Hospital, Kathmandu, Nepal for 1 year. All newly admitted adult patients ≥ 16 years of age, expected to stay in ICU / critical care areas for at least 7 days, barring the exclusion criteria, will be included in the study and evaluated for MRC sum score and skeletal muscle thickness, echogenicity and fasciculations using ultrasound on day 1, day 4 and day 7. The measurements will then be statistically analyzed to see if there is any relationship between trend of changes in muscle thickness, echogenicity and fasciculations and ICU-AW

DETAILED DESCRIPTION:
All newly admitted patients (shifted to ICU within 48 h of hospital admission), aged ≥ 16 years and expected to stay in ICU or critical care areas for 7 days will be included in the study after excluding those who fulfill excluding criterial. In all the participants, muscle strength will be assessed at day 1, day 4 and day 7, if the patients are awake as assessed by Richmond Agitation Sedation Scale (RASS) (19) between -1 and 1, and cooperative (20) assessed by being able to follow at least 3 out of 5 verbal commands with facial muscles (scored by the Score of 5 Questions). Assessment will be done by an ICU physician blinded to the result of ultrasound. The MRC score will be used for assessment of strength in the following six muscle groups bilaterally: wrist dorsiflexors, elbow flexors, shoulder abductors, hip flexors, knee extensors and ankle dorsiflexors. ICU-AW will be defined as MRC sum score < 48, in accordance with the international consensus statement.(1) Muscle ultrasound measurements (the index test) Muscle ultrasound will be performed by an ICU faculty or a DM resident of Critical care medicine (who has an experience of at least 25 muscle ultrasonography with at least 10 muscle ultrasonography performed under supervision) (21) and will be blinded to the result of MRC score of the patient. Muscle ultrasound images on day 1, day 4 and day 7 will be obtained in the participants, using Mindray DC-60® portable ultrasound machine, with a 9 to 13 MHz linear probe. The device settings include MSK pre-set, and will be kept constant during all examinations. The depth can be altered individually when deeper view is required to visualize the entire muscle thickness. Patients will be examined in the supine position with extended upper, lower limbs and completely relaxed muscles. The relaxation of muscle will be ensured by scanning the muscle in the sagittal view. A contracted muscle will show bulging in the central portion with thinning of its more distal ends. The angle of pennation can be seen to change as the muscle moves through its range of motion and the interosseous membrane will show bulging. A generous amount of contact gel will be used to minimize the required pressure of the transducer on the skin. Compression of the tissue will be avoided as it can affect the quality of muscle images. Transverse images of each muscle will be obtained with the transducer perpendicular to the direction of muscle fibre orientation.

The following parameters will be measured by muscle ultrasound

1. Muscle thickness
2. Muscle echogenicity
3. Muscle fasciculations Muscle thickness Measurements will be made using the built-in electronic calipers on a frozen, real time, cross section image over the largest bulk visible to eye. 3 measurements will be taken at each site and the mean value used for statistical analysis. The following anatomical sites will be assessed bilaterally: (22)

   * The biceps brachii muscle including the underlying brachialis muscle
   * The forearm flexor group
   * The quadriceps femoris muscle
   * The tibialis anterior muscle Muscle echogenicity The muscle echogenicity will be assessed by muscle ultrasound and graded according to Heckmatt and colleagues into four grades:(16) Grade I: Normal echo intensity with starry-night aspect with distinct bone echo.

Grade II: Increased echo intensity with normal bone echo. Grade III: Increased echo intensity with reduced bone signal. Grade IV: Increased echo intensity and loss of bone signal Muscle fasciculations The muscle fasciculations will be detected by ultrasound.(18) Each muscle will be examined over a time period of 10 seconds. The movement of fasciculation will be defined as twitching of small parts of the muscle lasting for 0.2-0.5 s, at least two of which will be required to be classified as being present. A fasciculation score ranges from 0 to 4 which is the number of regions with fasciculations out of four muscle regions. All the participants will be managed according to the ICU protocol of TUTH and there will be no variation in treatment between those allocated to study and those not allocated to the study.

ELIGIBILITY:
Inclusion Criteria:

* All newly admitted patients (shifted to ICU within 48 h of hospital admission)

  * Age ≥ 16 years
  * Expected to stay in ICU or critical care areas for 7 days

Exclusion Criteria:

* Patients with an admission diagnosis of a neuromuscular disorder

  * Patients with an admission diagnosis of stroke
  * Patients with an admission diagnosis of cardiac arrest
  * Patients with an admission diagnosis of traumatic brain injury
  * Patients with an admission diagnosis of spinal injury
  * Patients with an admission diagnosis of intracerebral infection or space-occupying lesion
  * Patients transferred from ICU of another hospital
  * Patients with a poor pre-hospital functional status (modified Rankin >3)
  * Patients in whom no arms or no legs were available for muscle strength testing or ultrasound

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly admitted adult patients ≥ 16 years of age expected to stay in ICU / critical care areas for at least 7 days
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the relationship between trend of changes in muscle thickness, echogenicity and fasciculations and ICU-AW among critically ill patients | 7 DAYS

CONTACTS AND LOCATIONS:
Overall Officials: MOHAN SHARMA, MBBS, MD, Mch, Study Director — IOM, TUTH, MMC
Locations (1):
- Institute of Medicine, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided